CLINICAL TRIAL: NCT05770466
Title: A Multicenter, Open-label, Randomized Study to Evaluate the Efficacy and Safety of Ropeginterferon Alfa-2b in the Treatment of Patients With Moderate COVID-19
Brief Title: Clinical Study for the Efficacy and Safety of Ropeginterferon Alfa-2b in Moderate COVID19.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202108013MIPC
Record Dates: First submitted 2022-07-14; First posted 2023-03-15 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Treated with P1101 (Ropeginterferon alfa-2b) plus standard of care (SOC)
  Interventions: Drug: P1101 (Ropeginterferon alfa-2b); Procedure: SOC
- Control group (Active Comparator): Treated with SOC alone
  Interventions: Procedure: SOC

INTERVENTIONS:
Drug: P1101 (Ropeginterferon alfa-2b) — 1. Name: P1101 (Ropeginterferon alfa-2b)
  2. Dosage form: pre-filled syringe
  3. Strength: A single dose of 250 mcg/0.5 mL
  4. Dosage and administration: 250 mcg per subcutaneous injection
  5. Mechanism of action (if known): Interferon work by binding to specific membrane receptors on the cell surface which in turn induce a complex sequence of intracellular events. These events include the induction of particular enzymes, suppression of cell proliferation, inhibition of virus replication in virus infected cells and immunomodulating activities.
  6. Pharmacological category: Antineoplastic and immunomodulating agents/ Immunostimulants/ Cytokines
  Arms: Experimental group
Procedure: SOC — SOC includes infection prevention and control measures, supportive care, dexamethasone, and antiviral agents. The SOC is based on the Taiwan Centers for Disease Control (CDC) guidance and investigator's discretion.

SUMMARY:
To evaluate the efficacy of subcutaneous ropeginterferon alfa 2b ( P1101combined with standard of care (SOC) compared with standard care alone in hospitalized adults with moderate COVID 19.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to comprehend and willingness to provide a written ICF before enter the study;
2. Male or non-pregnant female patients, ≥ 20 years of age at the time of enrolment;
3. Hospitalized patient with a diagnosis of COVID-19 on the basis of a positive# reverse transcriptase polymerase chain reaction (RT-PCR) with moderate## disease on admission###. #: Ct value <30. ##:Disease severity as defined by the treatment guidance of Taiwan Centers for Disease Control (CDC):

   > Moderate: Pneumonia patients without severe symptoms, blood oxygen saturation ≥93% without supplemental oxygen equipment (on room air); ###: Confirmed positive RT-PCR result ≤ 4 days prior to screening visit is eligible
4. Agrees to the collection of pharyngeal swabs and blood sample as per protocol.

Exclusion Criteria:

1. Known history or presence of decompensated cirrhosis of the liver (Child-Pugh B or C) before study entry.
2. Patients with intubation, respiratory failure, septic shock, multiple organ dysfunction or need additional organ support (e.g. vasopressors or ECMO).
3. Patients who have SpO2 <93% on room air, respiratory frequency >30 breaths/min.
4. Patients treated by dexamethasone before Day 1.
5. Patients treated by supplemental oxygen (FiO2 >40%) before Day 1.
6. Stage ≥4 severe chronic kidney disease or requiring dialysis (i.e. eGFR <15 mL/min/1.73 m2).
7. Females who are breast-feeding, lactating, pregnant or intending to become pregnant.
8. Known history of severe allergic or hypersensitivity reactions, e.g. hypersensitivity to the active substance or to any of the excipients of ropeginterferon alfa-2b.
9. Known history or presence of poorly controlled or clinically significant medical conditions that are not suitable to be enrolled, at the discretion of the investigator: major psychiatric (including but not limited to those with severe depression, severe bipolar disorder, schizophrenia, suicidal ideation or history of suicidal attempt).

11. Clinically significant medical conditions known to interfere with absorption, distribution, metabolism or excretion of the study drugs.

12. Patients treated by monotherapy of telbivudine or any other combination therapy with telbivudine within 1 month prior to screening.

13.Therapy with any anti-neoplastic, or immunomodulatory treatment within 1 month prior to screening.

14. Patient who have been vaccinated with any live attenuated vaccine or COVID- 19 vaccine within 1 month prior to screening.

15. Use of an investigational medical product within 1 month prior to screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who are negative to SARS-CoV-2 at Day 8 | Up to Day 8
  Proportion of patients who are negative to SARS-CoV-2 based on quantitative (Ct value ≥30) RT-PCR at Day 8 or discharge before Day 8 due to recovery
Time to discharge from hospital | Up to Day 29
  Time to discharge from hospital according to the latest Taiwan CDC guidance for SARS-CoV-2 infection (From randomization to discharge)

SECONDARY OUTCOMES:
Proportion of patients who are negative to SARS-CoV-2 at Day 5 | Up to Day 5
  Proportion of patients who are negative to SARS-CoV-2 based on quantitative (Ct value ≥30) RT-PCR at Day 5 or discharge before Day 5 due to recovery
Change in clinical status of patient at Day 5 | Up to Day 5
  Change in clinical status of patient on WHO clinical progression scale at Day 5
Change in clinical status of patient at Day 8 | Up to Day 8
  Change in clinical status of patient on WHO clinical progression scale at Day 8
Change of SpO2 | Up to Day 29
  Change of SpO2 from baseline
Time from symptom onset to resolution of clinical signs and symptoms | Up to Day 29
  Time from the onset of clinical symptoms related to COVID-19 (e.g., fever, cough, dyspnea or change in taste or smell) to the resolution of clinical signs and symptoms.
Time from symptom onset to RT-PCR negative result | Up to Day 29
  Time from the onset of clinical symptoms related to COVID-19 (e.g., fever, cough, dyspnea or change in taste or smell) to the RT-PCR negative result (Ct value ≥30).
Time from RT-PCR positive result to the resolution of clinical signs and symptoms | Up to Day 29
  Time from RT-PCR positive result (Ct value < 30) to the resolution of clinical signs and symptoms related to COVID-19 (e.g., fever, cough, dyspnea or change in taste or smell)
Time from RT-PCR positive result to RT-PCR negative result | Up to Day 29
  Time from RT-PCR positive result (Ct value < 30) to RT-PCR negative result (Ct value ≥30)
Occurrence and duration (days) of supplemental oxygen | Up to Day 29
  Occurrence and duration (days) of supplemental oxygen
Occurrence and duration (days) of mechanical ventilation | Up to Day 29
  Occurrence and duration (days) of mechanical ventilation
Time to treatment with other antiviral agents within 8 days | Up to Day 8
  To evaluate the time to treatment with other antiviral agents within 8 days in the Ropeginterferon alfa-2b treatment group,

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No